CLINICAL TRIAL: NCT02046681
Title: Monitoring Side Effects Of Pain Medication Prescribing By Emergency Department In Patients Over 65. The MOSE65 Study
Brief Title: Monitoring Side Effects Of Pain Medication Prescribing By Emergency Department In Patients Over 65
Acronym: MOSE65
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera S. Maria della Misericordia (Other)
Responsible Party: Principal Investigator, Ciro Paolillo, Dr. Ciro Paolillo, Azienda Ospedaliera S. Maria della Misericordia
Other Study IDs: AOSMariaMisericordia
Record Dates: First submitted 2014-01-09; First posted 2014-01-28 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2014-06

CONDITIONS: Acute Pain; Analgesics; Elderly
Keywords: Medication Adherence; Medication Compliance; Medication Therapy Management; Side effects; Analgesics; Emergency Medicine; Home care; Aged; Acetaminophen; codeine; ibuprofen; Oxycodone
MeSH Terms: conditions — Acute Pain; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acetam, acetam + codeine, Ibuprofen, Oxycodone: monitoring side effects of pain medication prescribed in patients over 65 acetaminophen 1000 mg tabs po q6h acetaminophen + codeine 500 mg tabs po q6h ibuprofen 200 mg tabs po q8h oxycodone 5 mg tabs po bid

SUMMARY:
Half of the people over the age of 65 are not functioning at their optimal level because of interference from pain. > 50% of older adults had taken prescriptions of pain medication beyond a 6-month period. In Emergency Department 80% of visits involving conditions with painful component. The study aims to observe and check side effects of most frequently pain killers prescribing at home to patients over 65 years old after a visit in emergency department.

DETAILED DESCRIPTION:
- observe side effects of pain medications prescribed in emergency department to patient over 65 yo

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* new analgesic treatment po following emergency department visits
* easily reachable by phone

Exclusion Criteria:

* age under 65
* pt may not able to hear, or answer the phone
* pt with a history of dementia
* pt who already takes pain killer, or neuroleptics

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: individuals age 65 years or older initiating analgesic treatment po following emergency department visits.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
To measure side effects of pain medication prescribed by emergency department to patients older 65 years | up to 1 week
  To Measure the rate of mayor and minor complications and the number of hospitalization during the therapy

SECONDARY OUTCOMES:
To ascertain the number of patients pain free | 1 month
  July 1, 2014
Measure the number of patients that follow the therapy prescribed | 1 month
  July 1 2014

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Paolillo, Dr, Study Chair — AOU S.Maria della Misericordia Udine
Locations (5):
- Italy (5):
  - Emergency Department AOU S.Maria della Midericordia Udine, Udine, Udine
  - Castelfranco Veneto Emergency Department, Castelfranco Veneto
  - Dolo Emergency Department, Dolo
  - Mirano Emergency Department, Mirano
  - Montebelluna Emergency Department, Montebelluna